CLINICAL TRIAL: NCT01784458
Title: Observational Study of Relationship Between Intra-abdominal Hypertension and Severe Sepsis in Surgical Patients
Brief Title: Clinical Significance of Intra-abdominal Hypertension in Surgical Patients With Severe Sepsis
Status: Completed | Type: Observational
Sponsor: University of Ulsan (Other)
Responsible Party: Principal Investigator, Kyu-Hyouck Kyoung, kyu-Hyouck Kyoung/clinical assistant professor, University of Ulsan
Other Study IDs: 2009-0004
Record Dates: First submitted 2013-02-03; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Bowel Perforation; Abscess; Leakage; Peritonitis; Pneumonia
Keywords: severe sepsis; intra-abdominal hypertension; intra-abdominal pressure
MeSH Terms: conditions — Intestinal Perforation; Abscess; Peritonitis; Pneumonia; Sepsis; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intra-abdominal hypertension(IAH): IAH group : patients developing IAH non-IAH group : patients without IAH

SUMMARY:
* Intra-abdominal pressure(IAP) is defined as a steady state pressure of the abdominal cavity
* many studies have proved IAP as a prognostic factor that elevated IAP influences hemodynamics and multiple organs dysfunction
* In previous studies, most of them was based on the septic patients of medical diseases. And it is rare about sepsis of surgical diseases such as traumatized or postoperative patients
* We hypothesized that intra-abdominal hypertension may affect clinical course such as length of stay of intensive care unit, weaning of mechanical ventilation, proceeding of enteral feeding and mortality
* Our study was aimed to investigate prevalence of IAH and risk factors and to analyze clinical course and prognosis influenced by IAH in surgical patients with severe sepsis

DETAILED DESCRIPTION:
* Inclusion criteria older than 18 diagnosed as severe sepsis agreed on informed consent
* Exclusion criteria refused to participate in the study traumatic injuries on urethra or bladder open abdomen status
* Definition of severe sepsis organ failure more than one organ with sepsis arterial blood lactate concentration of at least 4mmol/L hypotension with a systolic blood pressure lower than 90mmHg
* Definition of intra-abdominal hypertension intra-abdominal pressure more than 12mmHg
* Measurement of IAP measuring via three lument urinary catheter measuring after filling with 25ml normal saline measuring in supine position at level of mid-axillary line on iliac crest measuring three times a day during ICU stay

ELIGIBILITY:
Inclusion Criteria:

* older than 18-year
* agreed on informed consent
* diagnosed with severe sepsis

Exclusion Criteria:

* traumatic injuries on urethra or bladder
* open abdomen status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to surgical intensive care unit with severe sepsis
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
effects of intra-abdominal hypertension on clinical course and outcome in surgical patients with severe sepsis | within 60 days after admission in surgical intensive care unit
  length of ICU stay length of hospital stay ventilator free days effect on enteral feeding 28 day and 60 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Kyung Hong, Study Director — Division of Trauma and Surgical Critical Care, Department of Surgery, University of Ulsan College of Medicine, Asan Medical Center, Seoul, Korea

REFERENCES:
- [Background] Cheatham ML, Malbrain ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. II. Recommendations. Intensive Care Med. 2007 Jun;33(6):951-62. doi: 10.1007/s00134-007-0592-4. Epub 2007 Mar 22. PMID 17377769
- [Background] Pelosi P, Croci M, Ravagnan I, Cerisara M, Vicardi P, Lissoni A, Gattinoni L. Respiratory system mechanics in sedated, paralyzed, morbidly obese patients. J Appl Physiol (1985). 1997 Mar;82(3):811-8. doi: 10.1152/jappl.1997.82.3.811. PMID 9074968
- [Background] Hering R, Wrigge H, Vorwerk R, Brensing KA, Schroder S, Zinserling J, Hoeft A, Spiegel TV, Putensen C. The effects of prone positioning on intraabdominal pressure and cardiovascular and renal function in patients with acute lung injury. Anesth Analg. 2001 May;92(5):1226-31. doi: 10.1097/00000539-200105000-00027. PMID 11323351
- [Background] Malbrain ML, Chiumello D, Pelosi P, Bihari D, Innes R, Ranieri VM, Del Turco M, Wilmer A, Brienza N, Malcangi V, Cohen J, Japiassu A, De Keulenaer BL, Daelemans R, Jacquet L, Laterre PF, Frank G, de Souza P, Cesana B, Gattinoni L. Incidence and prognosis of intraabdominal hypertension in a mixed population of critically ill patients: a multiple-center epidemiological study. Crit Care Med. 2005 Feb;33(2):315-22. doi: 10.1097/01.ccm.0000153408.09806.1b. PMID 15699833
- [Result] Malbrain ML, Cheatham ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Johansson K, Kolkman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. I. Definitions. Intensive Care Med. 2006 Nov;32(11):1722-32. doi: 10.1007/s00134-006-0349-5. Epub 2006 Sep 12. PMID 16967294
- [Derived] Kyoung KH, Hong SK. The duration of intra-abdominal hypertension strongly predicts outcomes for the critically ill surgical patients: a prospective observational study. World J Emerg Surg. 2015 May 30;10:22. doi: 10.1186/s13017-015-0016-7. eCollection 2015. PMID 26056530